CLINICAL TRIAL: NCT06933693
Title: Prevalence Effects in Visual Search: Theoretical and Practical Implications
Brief Title: Mixed Vs Blocked Search: Four Unique Tasks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Jeremy M Wolfe, PhD, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2007P000646-G; R01EY017001 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-21 (Actual); Status verified 2025-04

CONDITIONS: Vision; Healthy; Attention
Keywords: visual search; visual attention

STUDY DESIGN:
Intervention Model Description: Each observer will do 400 "mixed" trials and 400 "blocked trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blocked Trials (Experimental): There are four search tasks in this experiment. Each task will be presented in a separate block of 100 trials
  Interventions: Behavioral: Blocked Trials
- Mixed Trials (Experimental): There are four search tasks in this experiment. All tasks will be randomly mixed in a single block of 400 trials.
  Interventions: Behavioral: Mixed trials

INTERVENTIONS:
Behavioral: Mixed trials — All tasks will be randomly mixed in a single block of 400 trials.
  Arms: Mixed Trials
Behavioral: Blocked Trials — Each search task will be presented in a block of trials.
  Arms: Blocked Trials

SUMMARY:
The goal is to look for qualitative differences in visual search behavior when one search is performed many times in a row compared to when multiple search tasks are intermixed. Four search tasks are tested. In the Mixed condition, the four tasks are randomly changed from trial to trial. In the Blocked condition, each task is run as a block of 100 trials.

DETAILED DESCRIPTION:
NOTE: This registration is linked to a Human Subjects registration in ASSIST. That, in turn, is part of an NCI Grant, R01EY017001. The grant describes many proposed experiments and notes that many others might be done as follow-up studies. At the suggestion of the NIH, the investigators grouped these studies into several "studies", each covering multiple experiments. The experiment described here is part of Aim 1 of R01EY017001. It is not possible to register a set of experiments through the PRS system in CT.gov and it is not possible to file an annual report for the grant (RPPR) without an NCT number for projects that have started collecting participants. Accordingly, the investigators are describing one experiment here that would be part of the "Project 1" bundle of studies.

When scientists study visual search in the lab, they usually ask people to do dozens of instances of the same type of task in a block. (e.g., Please find a vertical line….in the next 100 trials). However, in many (maybe most) visual searches in the real world, the participants are rarely looking for the same item (or same type of item) back-to-back. You do one search. Then the participants do another, and so on. (Find the jam. Now, find the bread. Now find a knife, etc). We want to know if the investigators would get the same results if the investigators mixed different searches together as the investigators do when the investigators test in long blocks of one specific type of search. This is important because the investigators want to know if the rules, established by years of blocked experiments, continue to apply in the more mixed real world.

There are multiple variants of this mixed/block experiment. In Experiment 1, observers are trained on four different search tasks. Then they perform 400 trials in the Mixed condition and the Blocked condition. In the Mixed condition, the four tasks are randomly changed from trial to trial. In the Blocked condition, each task is run as a block of 100 trials. Stimuli are placed in random locations in a jiggled 5 x 5 grid. The grid are placed within square field that is 0.5 of the maximum height of the screen. Each stimulus item fit into an invisible box that is 0.11 of the screen height. If the viewing distance is about 60 cm, a standard computer screen would show a stimulus field of about 15 deg on a side and each item would be placed in a box of about 3 x 3 deg. The background is white. Trials are divided evenly between three set sizes: 8, 16, and 24 items and evenly between target-present and absent trials. Stimuli are presented until the observer responds by pressing either 'p' or 'q' to indicate target present or absent, respectively. Accuracy feedback is provided after each trial.

ELIGIBILITY:
Inclusion Criteria:

* Pass Ishihara color vision test

Exclusion Criteria:

* vision less than 20/25 with correction
* history of neuromuscular or visual disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Response Time (RT) | Through study completion, an average of one year
  How long it takes to respond that the target is present or absent.

SECONDARY OUTCOMES:
Accuracy | through study completion, an average of one year
  The rates of false positive and false negative errors

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Wolfe, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified information about age, sex, and individual data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be placed on the Open Science Framework (OSF) site and should be permanent
Access Criteria: open
URL: https://osf.io/26jsr